CLINICAL TRIAL: NCT06022029
Title: A Phase 1 Dose-Escalation and Expansion Study of Intratumorally Administered ONM-501 Alone and in Combination With Cemiplimab in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: A Dose Escalation and Dose Expansion Study of Intratumoral ONM-501 Alone and in Combination With Cemiplimab in Patients With Advanced Solid Tumors and Lymphomas.
Acronym: ON-5001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: OncoNano Medicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ON-5001
Record Dates: First submitted 2023-08-15; First posted 2023-09-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Triple Negative Breast Cancer; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Lymphoma, Non-Hodgkin; Mantle Cell Lymphoma; Bladder Cancer; Uveal Melanoma, Recurrent; Cervix Cancer; Carcinoma in Situ; Head and Neck Squamous Cell Carcinoma; Skin Cancer; Metastatic Cancer; Tumor, Solid; Tumor Recurrence
Keywords: Solid tumors; Lymphoma; ONM-501; STING; Intra-tumoral; HNSCC; Breast Cancer; Melanoma; Skin Cancer; cemiplimab; Libtayo; DLBCL; bladder cancer; cervical cancer; metastases; immunotherapy; ICI; TNBC; Triple Negative; mTNBC; anti-PD-1 antibody; BRCA1; BRCA2; anti-PD-L1; uveal; NHL; Mantle Zone lymphoma; FL; stimulator of interferon genes
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Urinary Bladder Neoplasms; Uveal Melanoma; Recurrence; Uterine Cervical Neoplasms; Carcinoma in Situ; Squamous Cell Carcinoma of Head and Neck; Skin Neoplasms; Neoplasm Metastasis; Neoplasms; Lymphoma; Bites and Stings; Breast Neoplasms; Melanoma | interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: In Part 1a patients will receive ONM-501 as a single agent; in Part 1b patients will receive ONM-501 in combination with Cemiplimab; Part 2 will be an expansion of ONM-501 in combination with Cemiplimab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1a: Monotherapy Dose Escalation (Experimental): ONM-501 will be administered as intratumoral injections once per week for three weeks, followed by three weeks without ONM-501 administration. Each dosing cycle will be 21 days.
  Interventions: Drug: ONM-501
- Part 1b: ONM-501 in Combination with cemiplimab (Experimental): ONM-501 will be administered as intratumoral injections once per week for three weeks followed by three weeks without ONM-501 administration. Each dosing cycle will be 21 days. The combination agent will be administered according to standard protocol, once every three weeks.
  Interventions: Drug: ONM-501; Drug: Cemiplimab
- Part 2: RDE ONM-501 in Combination with cemiplimab in indication-specific expansion cohorts (Experimental): Once the recommended doses for expansion (RDEs) are determined for ONM-501 + ICI combination or ONM-501 monotherapy, the expansion phase of the study will be initiated. The expansion phase will enroll patients in one to three indication-specific expansion cohorts.
  Interventions: Drug: ONM-501; Drug: Cemiplimab

INTERVENTIONS:
Drug: ONM-501 — Intratumoral injection
Drug: Cemiplimab — Intravenous administration of 350 mg
  Other Names: Libtayo
  Arms: Part 1b: ONM-501 in Combination with cemiplimab; Part 2: RDE ONM-501 in Combination with cemiplimab in indication-specific expansion cohorts

SUMMARY:
A phase 1, multicenter, open label, non-randomized dose escalation and dose expansion study to examine the maximum tolerated dose, (MTD), minimum effective dose (MED) and/or recommended dose for expansion (RDE) of intratumoral ONM-501 as monotherapy and in combination with a PD-1 checkpoint inhibitor in patients with advanced solid tumors and lymphomas.

DETAILED DESCRIPTION:
This Phase 1, multi-center trial will consist of three parts: monotherapy dose escalation; combination therapy dose finding; and combination therapy dose expansion exploring two doses in specific tumor indication(s). Each dosing cycle of ONM-501 will be 21 days. ONM 501 will be administered as intratumoral injections once per week for three weeks (on Days 1, 8, and 15), followed by three weeks without ONM-501 administration. The monotherapy dose escalation will utilize an accelerated titration method.

The combination agent will be administered according to standard protocol, once every three weeks. This phase will evaluate ONM-501 in combination with approved immune checkpoint inhibitor (ICI) cemiplimab. Enrollment in this phase will follow a "Rolling 6" or 6+0 methodology - up to 6 patients will be enrolled in a staggered format; dose escalation of ONM-501 will be permitted.

Once the recommended doses for expansion (RDEs) are determined for ONM-501 + ICI combination or ONM-501 monotherapy, the expansion phase of this study will be initiated. The expansion phase will enroll patients in one to three indication-specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign written informed consent before performance of any study procedures
2. Age ≥ 18 years
3. Participants with solid tumors or lymphomas, confirmed by available histopathology records or current biopsy, that are advanced, nonresectable, or recurrent and progressing since last antitumor therapy, and for which no alternative standard therapy exists.
4. Participants must have a minimum of one injectable and measurable lesion.
5. Participants with prior Hepatitis B or C are eligible if they have adequate liver function
6. Participants with human immunodeficiency virus (HIV) are eligible if on established HAART for a minimum of 4 weeks prior to enrollment, have an HIV viral load <400 copies/mL, and have CD4+ T-cell (CD4+) counts ≥ 350 cells/uL
7. Adequate bone marrow function:
8. Adequate liver function

Exclusion Criteria: Patients will be excluded from this study if they meet any of the following criteria (Part 1a and Part 1b).

1. Other malignancy active within the previous 2 years except for basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast that has completed curative therapy.
2. Major surgery within 4 weeks before the first dose of study drug.
3. Brain metastases that are untreated or in the posterior fossa or involve the meninges. Participants with stable or previously treated progressing brain metastases (except in the posterior fossa or involving the meninges) may be permitted in a case-by-case basis at the Sponsor's discretion.
4. Prolongation of corrected QT (QTc) interval to >470 millisecond (ms) for males and females when electrolytes balance is normal.
5. Females who are breastfeeding or pregnant at screening or baseline
6. Females of childbearing potential that refuse to use a highly effective method of contraception.
7. Has uncontrolled or poorly controlled hypertension as defined by a sustained BP > 9. Has received prior investigational therapy within 5 half-lives of the agent or 4 weeks before the first administration of study drug, whichever is shorter.
8. Has had any major cardiovascular event within 6 months prior to study drug 10. Has known hypersensitivity to any component in the formulation of ONM-501
9. Has an active infection requiring systemic treatment
10. Is participating in another therapeutic clinical trial

Additional Exclusion Criteria for ONM-501 in Combination with cemiplimab (Part 1b)

1. Has known hypersensitivity to any component in the formulation of cemiplimab
2. Has any active or recent history of a known or suspected autoimmune disease or recent history of a syndrome that required systemic corticosteroids (>10 mg daily prednisone equivalent)
3. Has a condition requiring systemic treatment with corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation and Expansion Phases: Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) and Based on TEAEs Severity | Up to approximately 24 months
  AE incidence will be coded using Medical Dictionary for Regulatory Activities (MedDRA) terminology. AE severity will be graded according to NCI CTCAE version 5.0 or later. Grade 1 scales as Mild (asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated); Grade 2 scales as Moderate (minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living [ADL]); Grade 3 scales as Severe (severe or medically significant but not immediately life threatening hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL); Grade 4 scales as Life-threatening consequences, urgent intervention indicated, and Grade 5 scales as Death related to Adverse Event (AE)
Dose Escalation and Expansion Phases: Number of Participants with Dose-Limiting Toxicities (DLTs) | Up to approximately 24 months
  DLT will be defined as the occurrence of any of the following events in the first 28 days of treatment in the dose escalation cohorts in Part 1 of the study or in the first 28 days of treatment for the first 6 patients at any dose in Part 1b (DLT observation periods). Any adverse event resulting in a dose hold or delay of ≥ 28 days will be considered a DLT. Toxicity will be evaluated according to NCI CTCAE version 5.0.
Dose Escalation and Expansion Phases: Number of Participants Reporting One or More Treatment Emergent Serious Adverse Event (SAEs) | Up to approximately 24 months
  AE incidence will be coded using Medical Dictionary for Regulatory Activities (MedDRA) terminology. AE severity will be graded according to NCI CTCAE version 5.0 or later.

SECONDARY OUTCOMES:
Dose Escalation and Expansion Phases: Cmax | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  Cmax is defined as the Maximum Observed Plasma Concentration for ONM-501
Dose Escalation and Expansion Phases: t1/2z | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  t1/2z is defined as the Terminal Disposition Phase Half-life for ONM-501
Dose Escalation and Expansion Phases: Tmax | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  Tmax is defined as the Time to Reach the Maximum Plasma Concentration (Cmax) for ONM-501
Dose Escalation and Expansion Phases: AUCt | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  AUCt is defined as the Area Under the Concentration-time Curve from Time 0 to Time t for ONM-501
Dose Escalation and Expansion Phases: AUCinf | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  AUCinf is defined as the Area Under the Concentration-time Curve from Time 0 to Infinity for ONM-501
Dose Escalation and Expansion Phases: CL/F | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  CL/F is defined as the apparent clearance of ONM-501 (CL/F), where F is the fraction of the dose absorbed.
Dose Escalation and Expansion Phases: Vz/F | Dose Escalation and Expansion Phases: Cycle 1 Day 1 and Cycle 1 Day 8 (each cycle is 21 days): predose and at multiple timepoints (up to 24 hours).
  Vz/F is defined as the apparent volume of distribution of ONM-501 (CL/F), where F is the fraction of the dose absorbed.
Expansion Phase Only: Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response will be defined as a best response of CR or PR. The objective response rate (ORR) will be calculated as the proportion of patients in the Efficacy Analysis Set who achieve an objective response. ORR will be assessed based on Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.
  Characterize the plasma pharmacokinetics (PK) of IT ONM-501 as monotherapy and in combination with cemiplimab
  Evaluate additional measures of clinical benefit including: Duration of Response (DOR), Progression Free Survival (PFS) by RECIST and Overall Survival
Expansion Phase Only: Duration of Response (DOR) | Up to approximately 24 months
  DOR analyses will be conducted for those patients in the Efficacy Analysis Set who achieve an objective response and is defined as the time from first objective status assessment of CR or PR until documentation of objective disease progression or death from any cause. Patients who do not progress and do not die will be censored on the date of last adequate tumor assessment. If no further adequate post-treatment tumor assessments were obtained for a patient, DOR will be censored at the date of the objective response (i.e., zero duration). DOR will be assessed based on RECIST v1.1.
Expansion Phase Only: Progression-Free Survival (PFS) | Up to approximately 24 months
  PFS is defined as the time from administration of the first dose of ONM-501 until documentation of objective disease progression or death from any cause. Patients who do not progress and do not die will be censored on the date of last adequate tumor assessment. If no adequate post treatment tumor assessments were obtained for a patient, PFS will be censored at Day 1 (i.e., zero duration). The PFS analysis will be conducted using the Safety Analysis Set.
  Assess the biological effects of IT ONM-501 demonstrated by changes in immune cells, immune cell markers, serum cytokines (such as TNF-⍺, IFN-⍺, IFN-β, and others consistent with activation of the cGAS-STING pathway) and gene expression patterns
Expansion Phase Only: Overall Survival (OS) | Up to approximately 24 months
  OS is defined as the time from the date of first dose administration to the date of death.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (9):
  - California Research Institute, Los Angeles, California
  - BRCR Global, Tamarac, Florida
  - Gabrail Cancer Center Research, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Australia (7):
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Cancer Care Wollongong, Wollongong, New South Wales
  - University of the Sunshine Coast Clinical Trials, Buderim, Queensland
  - Tasman Oncology Research, Southport, Queensland
  - Princess Alexandra Hospital | Metro South Health, Woolloongabba, Queensland
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia